CLINICAL TRIAL: NCT03435380
Title: EMPOWER-II: Promoting Breast Cancer Screening in Women Who Survived Childhood Cancer
Brief Title: Promoting Breast Cancer Screening in Women Who Survived Childhood Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); St. Jude Children's Research Hospital (Other); Memorial Sloan Kettering Cancer Center (Other); City University of New York, School of Public Health (Other); University of California, San Francisco (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00088926; R01CA134722 (NIH)
Record Dates: First submitted 2018-02-01; First posted 2018-02-19 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Breast Neoplasms; Early Detection of Cancer
Keywords: Cancer Survivors; Smartphone; Mobile Applications
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned, in a ratio of 1:1:1, to one of the three groups: control, patient activation (PA), or patient activation + primary care provider activation (PA+PCP). Participants will remain in the group they are randomized to with no crossover throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (C) (Experimental): Targeted mailed educational materials (C).
  Interventions: Behavioral: Control
- Patient activation (PA) (Experimental): C + patient activation (PA) consisting of (1) smartphone app with HIPAA compliant survivorship care plan that can be viewed, printed, or emailed to their primary care provider; and (2) two-way (interactive) tailored text messages with links to video vignettes discussing the primary barriers to breast MRI and mammography.
  Interventions: Behavioral: Patient activation; Behavioral: Control
- Patient activation + primary care provider activation (PA+PCP) (Active Comparator): C + PA + PCP activation (PA+PCP) with physician materials about breast cancer risk in this population along with national and international guidelines for breast cancer surveillance.
  Interventions: Behavioral: Patient activation; Behavioral: Primary care physician activation; Behavioral: Control

INTERVENTIONS:
Behavioral: Patient activation — Smartphone-based materials including text messages and supplemental short videos focusing on how to find a primary care doctor, the importance of medical screening, and how to talk to a doctor about medical screening. Guidelines for monitoring and maintaining health, such as a survivorship care plan, will also be included in the smartphone-based materials.
  Arms: Patient activation (PA); Patient activation + primary care provider activation (PA+PCP)
Behavioral: Primary care physician activation — Mailed educational print materials sent to the participants' primary care doctors about health risks and recommendations for medical screening for adult women who were treated for a childhood cancer with chest radiation.
  Arms: Patient activation + primary care provider activation (PA+PCP)
Behavioral: Control — Mailed educational materials.

SUMMARY:
The primary purpose of this study is to determine the impact of maximizing patient and primary care provider (PCP) activation on breast cancer surveillance rates among women previously treated with chest radiotherapy (RT) for a childhood cancer. This is an 18-month, 3-arm randomized controlled trial using a smartphone intervention with data being collected at baseline and 18-months through patient and provider surveys and medical record review. Eligible women treated for a childhood cancer with chest RT will be randomly sampled from the Childhood Cancer Survivor Study (CCSS) and randomly selected to one of three groups: control, patient activation (PA) using a smartphone-based intervention, or patient activation + primary care provider activation (PA+PCP) which will include physician materials about breast cancer risk in this population along with guidelines for breast cancer surveillance. Participants in all groups will receive mailed targeted print materials as an educational resource about their previous chest radiation and breast cancer screening recommendations. The primary outcome is a medical record confirmed breast MRI and mammogram with the goal of increasing the rate of women completing the national guideline-based recommended combination of breast MRI and mammogram. This study will test the hypothesis that women in the PA and PA+PCP groups will have significantly higher rates of breast cancer surveillance (breast MRI and mammogram) than women in the control group. In addition, the hypothesis that women in the PA+PCP group will have significantly higher rates of breast cancer surveillance than women in the PA group will also be tested.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will include women who:

* Were diagnosed with a childhood cancer prior to the age of 21 years;
* Were treated with ≥ 10 Gy of chest RT (recent revision with a lower dose threshold);1
* Do not have a history of breast cancer;
* Have not had both a breast MRI and mammogram in the previous 24 months;
* Do not have a contraindication to MRI (i.e., pacemaker);
* Are 25 years of age or older at time of enrollment;
* Have an interval from their chest RT to the time of enrollment of at least 8 years;
* Have a smartphone;
* Are English-speaking.

Participants will be selected from women in the Childhood cancer Survivor Study (CCSS) cohort.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Oeffinger, MD, Principal Investigator — Duke University; Jennifer S Ford, PhD, Principal Investigator — City University of New York, School of Public Health
Locations (5):
- United States (5):
  - Columbia University, New York, New York
  - Hunter College, City of New York, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
Participants will be recruited from an established cohort (Childhood Cancer Survivor Study), and therefore individual participant data will not be available to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 12 waves from 5/7/2019 to 12/1/2020. The CCSS Coordinating Center sent introductory letters of invitation via email, regular mail, or phone. Interested participants were then given instructions on how to download the Eureka app from which they completed an electronic consent form and HIPAA waiver. All recruitment and study activities were completed remotely through the Eureka app.
Pre-assignment Details: 43 participants did not complete the baseline survey for varying reasons and were not randomized.
Period: Overall Study
Arm/Group | Control (C) | Patient Activation (PA) | Patient Activation + Primary Care Provider Activation (PA+PCP)
Started | 90 | 91 | 90
Completed | 76 | 79 | 81
Not Completed | 14 | 12 | 9
Not completed — Death | 1 | 2 | 1
Not completed — Lost to Follow-up | 12 | 8 | 6
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Ineligible | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (C) | Patient Activation (PA) | Patient Activation + Primary Care Provider Activation (PA+PCP) | Total
Number analyzed (Participants) | 90 | 91 | 90 | 271
Age, Continuous [Median (Full Range); unit: years] | 42 [27 to 68] | 42 [28 to 68] | 42 [27 to 62] | 42 [27 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 91 | 90 | 271
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 7 | 12
  Not Hispanic or Latino | 83 | 90 | 79 | 252
  Unknown or Not Reported | 3 | 0 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 2 | 3
  Race: Asian or Other Pacific Islander | 2 | 1 | 0 | 3
  Race: Black or African American | 5 | 3 | 5 | 13
  Race: White | 80 | 85 | 81 | 246
  Race: Other | 2 | 1 | 2 | 5
  Race: Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90 | 91 | 90 | 271

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women Who Completed a Breast MRI and Mammogram
Description: Self-reported
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control (C) | Patient Activation (PA) | Patient Activation + Primary Care Provider Activation (PA+PCP)
Number analyzed (Participants) | 90 | 91 | 90
percentage of participants | 8.9 [4.6 to 16.6] | 22.0 [14.7 to 31.5] | 17.8 [11.2 to 27.0]
Statistical Analysis 1: Comparison: Control (C) vs Patient Activation (PA); Test type: Superiority; p = 0.019, Mantel Haenszel; Stratified by age at consent (25-39 vs >=40), diagnosis (Hodgkin lymphoma vs other) and previous breast imaging exam (either mammogram or breast MRI); Risk Ratio (RR) = 2.37, 95% CI 2-sided [1.11 to 5.07]
Statistical Analysis 2: Comparison: Control (C) vs Patient Activation + Primary Care Provider Activation (PA+PCP); Test type: Superiority; p = 0.092, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.96, 95% CI 2-sided [0.87 to 4.38]

2. Other Pre Specified Outcome: Patient Activation Measure (PAM) - Questionnaire
Description: Measures patient activation and includes: believing one has an active role to play, having the confidence and knowledge to take action, taking action, and staying the course under stress.
Time Frame: 18 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Breast Cancer Surveillance Practices - Knowledge of Recommendations (Questionnaire)
Description: The Breast Cancer Surveillance Practices instrument (questionnaire) was developed as part of an effort supported by NCI funding (R21CA106972) and published in JAMA (Oeffinger KC, et al. JAMA, 301:404-414, 2009). The section regarding knowledge of the recommendations was then adapted for the EMPOWER-I Study, supported by NCI R01134722, and includes 3 items to determine if participants have (1) heard of mammography for breast cancer screening (yes, no, not sure), at what age women like the participant should begin getting a mammogram, and how frequently (multiple time frames).
Time Frame: 18 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Barrier Scales (Questionnaire)
Description: Elicits a rank order of the most relevant and important barriers of breast MRI and those associated with mammogram, for those women who did not obtain the recommended screening. The barriers are presented as a list of 13 statements in which there are 5 ranges of measure provided for each statement. The scale ranges include "Not at all," "A little bit," "Moderately," "Quite a bit," and "Extremely." The value/response of "Not at all" is considered to be the better outcome, whereas the value/response of "Extremely" is considered to be the worst outcome for the barrier scale. The scale is not combined to compute a total score, since responses are scored for each statement individually.
Time Frame: 18 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Pros and Cons of Mammography and Breast MRI (Questionnaire)
Description: The Pros and Cons of mammography is a 13-item instrument developed by Rakowski et al (Prev Med 1997). It was used in our Breast Cancer Surveillance Practices instrument (Oeffinger KC, et al. JAMA, 2009). The pros and cons scores (5-point Likert items) are converted to T-scores and then presented as a summary Decisional Balance. For EMPOWER-I Study, we adapted this instrument to also assess a woman's perspective on the pros and cons of breast MRI. This resulted in a 7-item instrument that is analyzed similar to the Pros and Cons of Mammography and presented as a Decisional Balance.
Time Frame: 18 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Family History of Breast Cancer (Questionnaire)
Description: This one-item question asks participants whether their mother, sister(s), or daughter(s) have been diagnosed with breast cancer.
Time Frame: 18 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Perception of Breast Cancer Risk (Questionnaire)
Description: This item was developed for the aforementioned Breast Cancer Surveillance Practices instrument and is a one-time question with asking women how they estimate their risk of breast cancer (with five responses: much more than the average woman, more than the average woman, same as the average woman, less than the average woman, much less than the average woman).
Time Frame: 18 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Communication With PCP (Questionnaire)
Description: Developed for the EMPOWER-I study, the questionnaire asks participants at the end of the study whether they saw a health care provider during the 18-month study period, whether they discussed breast cancer screening with a provider, and whether the provider responded to the information (5-point Likert). Each of these items will be analyzed separately.
Time Frame: 18 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Affect
Description: Will be measured using the adapted and shortened version of the Positive Affect Negative Affect Scale (PANAS). We will focus on emotions related to managing health.
Time Frame: 18 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Future Breast Screening Intentions
Description: To determine the Stage of Adoption (Change) for breast cancer surveillance, participants will be asked when they plan to have their next mammogram and/or breast MRI (following the completion of the study).
Time Frame: 18 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Self-Efficacy
Description: Measures confidence in discussing breast surveillance with the primary care physician and obtaining the recommended screening using items developed by Champion and colleagues.
Time Frame: 18 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Primary Care Provider Demographics
Description: Age, gender, years in practice, and practice setting.
Time Frame: Baseline
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Primary Care Provider Experience
Description: Most PCPs have taken care of only a few childhood cancer survivors. To ascertain their past experience with caring for this population, we ask PCPs how many childhood cancer survivors they have in their practice panel (0, 1-2, 3-5, >5).
Time Frame: 18 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Primary Care Provider Comfort Level
Description: Comfort level with caring for adult survivors of childhood cancer (Likert scale)and familiarity with available guidelines (Likert scale).
Time Frame: 18 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Primary Care Provider Knowledge
Description: Using a hypothetical vignette of a 29-year old female patient treated for Hodgkin lymphoma with chemotherapy and chest RT, questions will be asked about screening for thyroid dysfunction, breast cancer, and cardiac dysfunction.
Time Frame: 18 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Economic Measurements
Description: Replication costs of the intervention and health services from the intervention per participant.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | Control (C) | Patient Activation (PA) | Patient Activation + Primary Care Provider Activation (PA+PCP)
All-Cause Mortality (participants affected / at risk) | 1/90 | 2/91 | 1/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/91 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/91 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT03435380/Prot_SAP_000.pdf